CLINICAL TRIAL: NCT02385435
Title: Comparison of Caudal Bupivacaine Alone With Bupivacaine Plus Two Doses of Dexmedetomidine for Postoperative Analgesia in Pediatric Patients Undergoing Infra-umbilical Surgery: A Randomized Controlled Double Blinded Study
Brief Title: Caudal Bupivacaine vs Bupivacaine Plus Two Doses of Dexmedetomidine for Postoperative Analgesia in Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Khaled Radian Al-zaben, Dr, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: University of jordan
Record Dates: First submitted 2015-02-24; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Pain, Postoperative
Keywords: caudal block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bupivacaine (Active Comparator): single shot caudal plain bupivacaine at a dose of 2mg/kg is used as a reference control drug.
  Interventions: Drug: Bupivacaine
- dexmedetomidine 1μg.kg-1 (Active Comparator): Single shot Caudal dexmedetomidine 1μg.kg-1 used as the second arm intervention
  Interventions: Drug: dexmedetomidine 1μg.kg-1
- dexmedetomidine 2μg.kg-1 (Active Comparator): Single shot Caudal dexmedetomidine 2 μg.kg-1 used as the second arm intervention
  Interventions: Drug: dexmedetomidine 2μg.kg-1

INTERVENTIONS:
Drug: Bupivacaine — Caudal Bupivacaine 2 mg/kg single shot
  Other Names: Broup B
  Arms: Bupivacaine
Drug: dexmedetomidine 1μg.kg-1 — Caudal dexmedetomidine 1μg.kg-1, single shot
  Other Names: Group BD1
  Arms: dexmedetomidine 1μg.kg-1
Drug: dexmedetomidine 2μg.kg-1 — Caudal dexmedetomidine 2μg.kg-1, single shot
  Other Names: Group BD2
  Arms: dexmedetomidine 2μg.kg-1

SUMMARY:
The aim of this prospective randomized double-blind study was to compare the analgesic efficacy and the side effects of two doses of dexmedetomidine (1 and 2 µg.kg-1) co-administered with bupivacaine with bupivacaine alone for caudal analgesia in children undergoing infra-umbilical surgery.

DETAILED DESCRIPTION:
* Quality assurance plan for data validation and registry: After Data was registered, it was reviewed by a second person who compared it to the Data in patient data collection forms.
* Data check: carried out using Statistical Package for the Social Sciences (SPSS) variable definition protocols. Also data were entered in EXCEL sheets for comparisons to guarantee consistency.
* Source data verification: Paper case report forms and medical records.
* Standard Operating Procedures to address registry operations and analysis activities: Eligible patients were recruited after obtaining consent. Data was collected by qualified personnel rained on the process. Data was entered into Excel sheets and SPSS programs and compared for consistency. Analysis of Data was carried out by a qualified statistician. Adverse events were reported as yes/no variables. Data of patients who had Change in management was omitted from analysis.
* Sample size assessment: Sample size was calculated to detect a 65% reduction in the analgesic requirement during the first 24 h from 75% in the bupivacaine group with α= 0.05 and β=0.80.
* Plan for missing data: Patients with missing Data were omitted from statistical analysis.
* Statistical analysis plan: carried out using International Business Machines (IBM) statistics 19.0 statistical package for windows. Data were compared using analysis of variance for continuous variables, Kruskal-Wallis test for ordinal, and chi square test for categorical ones. Post hoc analyses were carried out as appropriate.

ELIGIBILITY:
Inclusion criteria:

* Patients with American Society of Anesthesiologists (ASA) - I
* Scheduled for lower abdominal and perineal surgery
* Under general anesthesia

Exclusion criteria:

* history of developmental delay or mental retardation
* known or suspected coagulopathy or recent use of anticoagulant/antiplatelet drugs.
* known allergy to any of the study drugs.
* any signs of infection or congenital abnormalities at the site of the proposed caudal block

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic requirement | 24 hours
  The time from end of surgery to the first requirement of postoperative analgesia
Postoperative pain scores | 24 hours
Number of postoperative analgesia doses | 24 hours
  Number of paracetamol doses needed by each patient

SECONDARY OUTCOMES:
Postoperative sedation scores | 2 hours
  Level of sedation was recorded throughout the post-anesthesia care unit stay at 15-minute time intervals.
Sevoflurane concentration | intraoperative
  Sevoflurane concentration required to maintain Bispectral Index (BIS) monitor reading between 40 and 60%.
Blood pressure | intraoperative
  Intraoperative blood pressure readings
Heart Rate | intraoperative
  Intraoperative heart rate readings
Side effects of study drugs | 24 hours
  Any side effects of study drugs in the first 24 hours postoperative hours were recorded (nausea, Vomiting, urine retention, lower limb weakness and emesis).

CONTACTS AND LOCATIONS:
Overall Officials: khaled R Al-zaben, Principal Investigator — University of Jordan; Ibraheem Y Qudaisat, Study Director — University of Jordan

REFERENCES:
- [Background] Tong Y, Ren H, Ding X, Jin S, Chen Z, Li Q. Analgesic effect and adverse events of dexmedetomidine as additive for pediatric caudal anesthesia: a meta-analysis. Paediatr Anaesth. 2014 Dec;24(12):1224-30. doi: 10.1111/pan.12519. Epub 2014 Sep 9. PMID 25203847
- [Background] She YJ, Zhang ZY, Song XR. Caudal dexmedetomidine decreases the required concentration of levobupivacaine for caudal block in pediatric patients: a randomized trial. Paediatr Anaesth. 2013 Dec;23(12):1205-12. doi: 10.1111/pan.12278. Epub 2013 Oct 12. PMID 24383602
- [Background] Bharti N, Praveen R, Bala I. A dose-response study of caudal dexmedetomidine with ropivacaine in pediatric day care patients undergoing lower abdominal and perineal surgeries: a randomized controlled trial. Paediatr Anaesth. 2014 Nov;24(11):1158-63. doi: 10.1111/pan.12478. Epub 2014 Jul 12. PMID 25040840
- [Background] Saadawy I, Boker A, Elshahawy MA, Almazrooa A, Melibary S, Abdellatif AA, Afifi W. Effect of dexmedetomidine on the characteristics of bupivacaine in a caudal block in pediatrics. Acta Anaesthesiol Scand. 2009 Feb;53(2):251-6. doi: 10.1111/j.1399-6576.2008.01818.x. Epub 2008 Dec 6. PMID 19076110
- [Background] El-Hennawy AM, Abd-Elwahab AM, Abd-Elmaksoud AM, El-Ozairy HS, Boulis SR. Addition of clonidine or dexmedetomidine to bupivacaine prolongs caudal analgesia in children. Br J Anaesth. 2009 Aug;103(2):268-74. doi: 10.1093/bja/aep159. Epub 2009 Jun 18. PMID 19541679
- [Background] Findlow D, Aldridge LM, Doyle E. Comparison of caudal block using bupivacaine and ketamine with ilioinguinal nerve block for orchidopexy in children. Anaesthesia. 1997 Nov;52(11):1110-3. doi: 10.1111/j.1365-2044.1997.204-az0346.x. PMID 9404178
- [Background] Xiang Q, Huang DY, Zhao YL, Wang GH, Liu YX, Zhong L, Luo T. Caudal dexmedetomidine combined with bupivacaine inhibit the response to hernial sac traction in children undergoing inguinal hernia repair. Br J Anaesth. 2013 Mar;110(3):420-4. doi: 10.1093/bja/aes385. Epub 2012 Nov 15. PMID 23161357
- [Background] Konakci S, Adanir T, Yilmaz G, Rezanko T. The efficacy and neurotoxicity of dexmedetomidine administered via the epidural route. Eur J Anaesthesiol. 2008 May;25(5):403-9. doi: 10.1017/S0265021507003079. Epub 2007 Dec 19. PMID 18088445
- [Background] Wu HH, Wang HT, Jin JJ, Cui GB, Zhou KC, Chen Y, Chen GZ, Dong YL, Wang W. Does dexmedetomidine as a neuraxial adjuvant facilitate better anesthesia and analgesia? A systematic review and meta-analysis. PLoS One. 2014 Mar 26;9(3):e93114. doi: 10.1371/journal.pone.0093114. eCollection 2014. PMID 24671181